CLINICAL TRIAL: NCT05411302
Title: Augmenting Mental Health Support for Patients Accessing Different Degrees of Formal Psychiatric Care Through a Supportive Text Messaging Program: A Randomized Controlled Trial
Brief Title: Augmenting Mental Health Support Through a Supportive Text Messaging Program
Acronym: Text4Support
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vincent Agyapong (Other)
Collaborators: Dalhousie University (Other); Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Vincent Agyapong, Psychiatrist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: Text4Support-NS47476
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Major Depressive Disorder; Generalized Anxiety Disorder; Mental Health Wellness 1
Keywords: Mental Health; Text messages; e-health; Text4Support
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Administrative data outcome assessors will be blinded to treatment group allocation by not involving them in discussions about study participants and not granting them access to the randomization code database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text4Support Arm (Experimental): Patients in the intervention (Text4Support) arm of the study will receive the usual care (i.e. community care, follow-up appointments), plus daily automated supportive text messages from an online application.
  Interventions: Other: Mental health supportive text messages
- Care as usual arm (No Intervention): Patients in the control arm of the study will receive the usual care, which includes the freely accessible Health Authority approved low-intensity e-mental health services. They will receive a single text message informing and encouraging them to utilize current MHAP resources on the NS Health website. They will not receive automated daily supportive text messages.

INTERVENTIONS:
Other: Mental health supportive text messages — Text4Support program was developed based on knowledge from randomized controlled trials conducted in Ireland and Alberta and from evaluations of the Text4Mood program. The diagnostic-specific approach is based on an analysis of service data, which suggested that diagnostic clusters for individuals accessing mental health services into 6 categories: mood disorders, anxiety disorders, schizophrenia and other psychotic disorders, substance use disorders, adjustment disorders and personality disorders. Thus, text message content will focus on 2 dimensions. General range includes messages of self-care, social support, hope, affirmation, and recovery. Specific content will focus on managing symptoms related to the conditions described above. As a component of scalability and inclusiveness, text message content can also be customized based on end-user characteristics. We will explore content that is sensitive to needs based on age group, cultural identity and gender identity.
  Arms: Text4Support Arm

SUMMARY:
Patients seeking mental health care and those being discharged from psychiatric units frequently express psychological distress. A lack of routine follow-up and tailored support during these critical stages of a patient's journey can weaken the patient's connection to the health care system, resulting in low adherence and dissatisfaction with treatment, and the need for more intensive therapies. These unfavourable outcomes may result in deterioration of the patient's mental health, readmissions, recurrent emergency department (ED) visits, and extended length of stay (LOS). The investigators propose implementing an add-on supportive text messaging service (Text4Support), developed using cognitive-behavioural therapy (CBT) principles to augment mental health support for patients accessing different degrees of psychiatric care in Nova Scotia. The primary objective is to investigate the effectiveness of Text4Support, compared to usual care, in improving clinical mental health outcomes and overall mental wellbeing among participants. Secondary objective is to examine the impact of Text4Support on health services utilization and patient satisfaction. Lastly, investigators will explore Text4Support implementation outcomes. This will be a multicenter, mixed-methods, longitudinal, prospective, parallel, two-arm, rater-blinded randomized controlled trial. Participants will be randomized into two arms: the intervention arm will receive the usual care, plus daily automated supportive text messages from an online application, and the control arm will receive the usual care, which includes the freely accessible Health Authority approved e-mental health services. It is planned to enrol at least 1500 participants. Quantitative data will be analyzed using repeated measures mixed-effects modelling, effect size analysis, and correlational analysis between measures at each time point on an intention-to-treat basis. Qualitative data analysis will be guided by the six-phase thematic analysis framework. The analysis of the implementation outcomes will be guided by the RE-AIM framework. The results of the study will provide important information with respect to a comprehensive evaluation of outcomes of a supportive daily text message program; comparability of a supportive daily text message program compared with care as usual; and the impact of a supportive daily text message program on clinical outcomes, patient satisfaction and health services utilization.

DETAILED DESCRIPTION:
In this study, the investigators are testing the Text4Support program, which is a daily supportive text message intervention, developed using cognitive-behavioural therapy (CBT) principles. The Text4Support program will be implemented in Nova Scotia/Canada, to augment mental health support for patients accessing different degrees of psychiatric care in the province.

The main goal is to evaluate how patients participating in community mental health programs or being discharged from psychiatric units will progress in terms of mental well-being and health services utilization if they receive daily automated supportive text messages from an online application, plus the usual care (i.e. community care, follow-up appointments). The results of this evaluation will be compared to the results from the patients who receive the usual care only. The prediction is that daily supportive text messages will result in a 20% greater reduction in the mean Patient Health Questionnaire 9 (PHQ-9), Generalized Anxiety Disorder 7 (GAD-7) scale, and Columbia Suicidal Rating Scale (CSRS) scores and a 20% greater increase in the Recovery Assessment Scale (RAS) and the World Health Organization 5 (WHO 5) Well-Being Index scores at 6 weeks, 3, 6 and 12 months from baseline compared to control interventions. It is also expected a reduction of 10-25% in services utilization (i.e. psychiatric readmissions and ED visits) among participants of the Text4Support arm, compared to the usual care group.

The length of this study for participants is 12 months. The entire study is expected to take about 3 years to complete. Results of this study are expected to be available within 3 years of project commencement. It is anticipated that about 1500 people will participate in this study throughout all zones of Nova Scotia.

Study procedures will include the following steps:

Screening:

A designated person from the patient's circle of care will provide a weekly list of potential participants (i.e., new patients enrolled in the TMHP, DH, RASP or MHCC, or patients expected to be discharged from the ED or PIU) to the research team, who will confirm eligibility before approaching the patients.

Informed consent process:

Patients enrolled in the TMHP, DH, RASP, or MHCC be provided with information about the study and facilitated on the day of program enrollment to complete the consent forms. Patients who are being discharged from the ED or PIU will be approached before leaving the unit. During the informed consent process, patients (and/or their parents/guardians, in the case of patients below 18 years old) will receive detailed information about the study's goal and procedures, risks and benefits, and participation alternatives. They can opt-in or opt-out of their participation in the RCT and/or the qualitative sub-study by providing consent or not. Participants will be advised about the voluntary nature of the study and that they may withdraw from the study at any time they want, without giving a reason. When a participant withdraws, no new health information will be gathered after that date. Information that was gathered before withdrawal may continue to be used if the participant agrees with that, otherwise, they can opt for full data withdrawal. Randomization and data collection will only be done after consent is obtained.

Randomization and Allocation:

The randomization process will use permuted blocks to ensure balance (1:1) between the two intervention groups. Patients will be randomized into one of two groups, namely, "Intervention Group" or "Control Group". Simple random allocation using a random number generator will be conducted by the research associate in order to ensure allocation concealment. The researcher who assigns patients to groups and sends text messages will not be involved in the baseline and follow-up assessments.

Blinding: As participants will be aware of whether or not they were receiving supportive text messages, blinding patients to their allocated experimental condition will not be possible. Administrative data outcome assessors will be blinded to treatment group allocation by not involving them in discussions about study participants and not granting them access to the randomization code database.

Individual interviews and focus groups:

A sub-sample from the overall pool of study participants will be drawn and invited by research team members to participate in the qualitative component of the study, which should be happening at the end of Quarter 2/Year 2. Inclusion criteria to take part in the qualitative sub-study are having previously provided consent and being available to attend a 2-hour, audio-recorded, individual interview and focus group session. Although the sub-sample will be drawn, both sex and gender-based representation will be considered in the sample, ensuring that at least ten non-male persons are included, as men are often over-represented in research. Investigators will also guarantee that different age groups, and those of marginalized groups are represented in this sample. The encounters will be conducted by a trained research team member in person or via Zoom. The focus group will have a maximum of 10 participants and last less than 1.5 hours. Participants will be offered a $40 gift card stipend during the enrollment process to thank them for their time and involvement.

As stated earlier, research participants will be randomized to one of the two groups named the Intervention Group and the Control Group, as detailed below:

The Intervention group:

Participants randomized to the intervention group will receive the usual care plus Text4Support. Usual care will comprise the standard care offered by each program/unit participating in this study (i.e. follow-up appointments or offering of community clinic/program treatment options). Text4Support will be provided through ResilienceNHope, which is an online application (https://application.resiliencenhope.com/) and offered by the Global Psychological eHealth Foundation (https://www.gpehealth.org/). Starting a day after enrolment, intervention-group participants will receive daily unidirectional (no-reply) supportive text messages for 12 months. The message content was created by psychiatrists, mental health therapists and mental health services users and is crafted based on cognitive behavioral therapy principles to address eight common mental health presentations and general wellbeing. Thus, automated daily text messages will consist of condition-specific symptom management content (eg, activity scheduling in depression, the importance of medication adherence) and general, widely indicated and symptomatology-independent content (eg, self-care, social support, hope, affirmation, and recovery content).

The Text4Support program was developed based on knowledge from randomized controlled trials conducted in Ireland and Alberta as well as from evaluations of the Text4Mood program in Alberta. Determination of a diagnostic-specific approach was based on an analysis of service data, which suggested that diagnostic clusters for individuals accessing Mental Health and Addiction services fell into six major categories: mood disorders, anxiety disorders, schizophrenia and other psychotic disorders, substance use disorders, adjustment disorders and personality disorders. Thus, text message content will focus on two dimensions. First, general content that is indicated regardless of symptomatology will be presented, including messages of self-care, social support, hope, affirmation, and recovery. Second, specific content will focus on the management of symptoms related to the specific conditions described above (e.g., activity scheduling in depression). As a component of scalability and inclusiveness, text message content can also be customized based on end-user characteristics. Specifically, investigators will explore content that is sensitive to needs based on age group, cultural identity and gender identity. This serves to enhance access for diverse groups, many of whom may be marginalized or underserved. If they wish to end their participation, subscribers just text "stop" and the messages stop; they receive this instruction as part of the welcome message.

The Control Group:

The control arm of the study will consist of usual care, which includes the follow-up appointments and/or offering of community clinic/program treatment options and the freely accessible Health Authority approved low-intensity e-mental health services. They will receive a single text message with the link to the MHAP open-access, and internet-based mental health resources, which are available at the website (https://mha.nshealth.ca/en/tools). Currently, there are 22 online tools available, covering a wide range of psychiatric conditions (i.e., substance abuse disorders, gambling, depression, anxiety, grief, bipolar disorders, eating disorders, obsessive-compulsive disorder, post-traumatic stress disorder, schizophrenia, psychosis, among others), group ages (children, youth, adult, seniors) and group identities (Black/African Nova Scotians, 2SLGBTQIA+, Canadian Forces, RCMP, Caregivers and families, First Nations/Indigenous people and first responders).

After providing consent and being assigned to one of the two study groups, participants will be officially enrolled in the study.

Research participants will be asked to do the following:

* Complete four (4) online questionnaires about mental health at enrollment, and 6 weeks, 3, 6, and 12 months after enrollment. The questionnaires will usually take a total of about 5 to 10 minutes to complete.
* Complete one (1) online questionnaire about satisfaction with the services they receive at 6 weeks, 3, 6, and 12 months after enrollment. This questionnaire will usually take a total of about 5 minutes to complete.
* Participants may be invited to an individual interview with researchers. The interview will be audio-recorded and may be in person or via Zoom, and will last about 30 minutes.
* During the interview, researchers will ask questions about patients' satisfaction and experience with the interventions received in the study.
* Participants may be invited to a group meeting with researchers and other participants in the study. This meeting is called a focus group interview. The encounter will be conducted by a trained research team member in person or via Zoom. The focus group will have a maximum of 10 participants and last about 1.5 hours, and the subject will be the participants' satisfaction and experience with the study interventions.

The link to the online surveys will be sent to the participants' mobile phones by text message. The link will be sent again if the participant does not complete the online surveys within a week of getting it. A research team member may call the participants to remind them to finish the questionnaires.

At the end of the study, participants can continue receiving the study intervention (Text4Support) after completing 12 months of research participation. Research participants may stop receiving text messages simply by texting "STOP" and the software will no longer send them text messages. This action can be done at any time during the study (i.e. if the patient wishes to withdraw from the study). The usual care will continue to be provided to all subjects after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Being a new patient (i.e. first-time user) of the TMHP, DH, RASP or MHCC, OR being a patient discharged from the ED or PIU (i.e. within a week period before discharge date).
* Ownership of a mobile device capable of receiving text messages.
* Able to read English text messages.
* Can provide informed written consent.

Exclusion Criteria:

* Patients who are not capable of reading text messages in English.
* Patients who are not own a mobile phone capable of receiving text messages.
* Patients who are not able/willing to provide consent to take part in the study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Well-being | Baseline, 6 weeks, 3, 6 and 12 months
  Change from Baseline to 6 weeks, 3, 6 and 12 months for the mean scores for the quality life, assessed through the World Health Organization 5 Well-Being Index (WHO-5) in both groups. WHO-5-Well-Being Index is a short 5-item generic global rating scale measuring subjective well-being. The scale was derived from the WHO-10, which in turn was derived from a 28-item rating scale. The scale has adequate validity both as a screening tool for depression and as an outcome measure in clinical trials. The raw score is calculated by totaling the figures of the five answers. The raw score ranges from 0 (zero) to 25, 0 (zero) representing worst possible and 25 representing best possible quality of life.To obtain a percentage score ranging from 0 to 100, the raw score is multiplied by 4. A percentage score of 0 (zero) represents worst possible, whereas a score of 100 represents best possible quality of life.
Change in Recovery | Baseline, 6 weeks, 3, 6 and 12 months
  Change from Baseline to 6 weeks, 3, 6 and 12 months for the mean scores for recovery, assessed through the Recovery Assessment Scale (RAS), in both groups. RAS is a 20-item measure developed based on a process model of recovery. The RAS evaluates various aspects of recovery with a special focus on hope and self-determination.
Change in Major Depressive Disorder | Baseline, 6 weeks, 3, 6 and 12 months
  Change from Baseline to 6 weeks, 3, 6 and 12 months for the mean scores for moderate to high depression (likely Major Depressive Disorder) assessed through the Patient Health Questionnaire (PHQ-9), in both groups. The PHQ-9 is a 9-item validated instrument used to diagnose and measure the severity of depression in general medical and mental health settings. PHQ-9 scores are: 0 - 4 None-minimal (patient may not need depression treatment); 5 - 9 Mild (use clinical judgment about treatment, based on patient's duration of symptoms and functional impairment); 10 - 14 Moderate (use clinical judgment about treatment, based on patient's duration of symptoms and functional impairment); 15 - 19 Moderately severe (treat using antidepressants, psychotherapy or a combination of treatment); 20 - 27 Severe (treat using antidepressants with or without psychotherapy).
Change in Generalized Anxiety Disorder | Baseline, 6 weeks, 3, 6 and 12 months
  Change from Baseline to 6 weeks, 3, 6 and 12 months in prevalence for moderate to high anxiety (likely Generalized Anxiety Disorder), assessed through the Generalized Anxiety Disorder (GAD-7) scale, in both groups. GAD-7 is a validated 7-item questionnaire used to assess the self-reported levels of anxiety in respondents. This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety; 15-21: severe anxiety.
Change in Suicidal Ideation and Behaviour | Baseline, 6 weeks, 3, 6 and 12 months
  Change from Baseline to 6 weeks, 3, 6 and 12 months in the mean score for suicidal ideation and behaviour, assessed through the Columbia-Suicide Severity Rating Scale, in both groups. C-SSRS is an assessment tool that evaluates suicidal ideation and behavior. The two initial questions have binary responses (yes/no), which lead to 10 different categories: 1) Wish to be Dead; 2) Non-specific Active Suicidal Thoughts; 3) Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; 4) Active Suicidal Ideation with Some Intent to Act, without Specific Plan; 5) Active Suicidal Ideation with Specific Plan and Intent; 6) Preparatory Acts or Behavior; 7) Aborted Attempt; 8) Interrupted Attempt; 9) Actual Attempt (non-fatal); 10) Completed suicide.

SECONDARY OUTCOMES:
Health services utilization (crisis calls) | 12 months
  Differences in health services utilization data (crisis calls), between groups.
Health services utilization (Emergency Department visits) | 12 months
  Differences in health services utilization data (ED visits) between groups
Health services utilization (hospital admissions) | 12 months
  Differences in health services utilization data (hospital admissions) between groups.
Health services utilization (hospital readmissions - i.e. admissions before 30 days os the last admission) | 12 months
  Differences in health services utilization data (readmissions) between groups.
Health services utilization (lenght of stay - LOS) | 12 months
  Differences in health services utilization data (LOS following inpatient hospitalization) between groups
Patient retention | 12 months
  Differences between groups of self-reported retention rates assessed through a 5-point Likert scale on the frequency of reading messages and returning to messages, and actions taken.
Patient satisfaction | 12 months
  Differences between groups of overall patient satisfaction using a 5-point self-designed Likert scale.

OTHER OUTCOMES:
Implementation (reach) | 6 weeks, 3, 6 and 12 months after enrollment
  Reach of the interventions will be assessed in the intervention group only, through administrative data about the proportion of target population who receive the daily supportive text messages across Nova Scotia.
Implementation (acceptability) | 12 months after enrollment
  Acceptability of the intervention will be assessed in the intervention group only, through instrument developed and pilot tested, and published by the authors.
Implementation (appropriateness) | 6 months after enrollment
  Appropriateness of the intervention will be assessed through qualitative in-depth individual interview.
Implementation (fidelity) | 6 weeks, 3, 6 and 12 months.
  Fidelity of the intervention will be assessed through administrative data about Percentage of participants who received text messages as planned (no technical issues).
Implementation (cost-effectiveness) | 6 weeks, 3, 6 and 12 months.
  Cost-effectiveness of the intervention, evaluated through adminstrative data about the incremental cost-effectiveness ratio (ICER) is the ratio between the difference in costs and the difference in benefits of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health - Abbie J. Lane Memorial Building QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Obuobi-Donkor G, Shalaby R, Agyapong B, Nkrumah SO, Adu MK, Eboreime E, Wozney L, Agyapong VIO. Impact of a supportive text messaging program (Text4Support) for mitigating psychological problems in patients receiving formal mental health services: A randomized controlled trial. Digit Health. 2025 Jul 23;11:20552076251361236. doi: 10.1177/20552076251361236. eCollection 2025 Jan-Dec. PMID 40727620